CLINICAL TRIAL: NCT02918409
Title: IV Colistin for Pulmonary Exacerbations: Improving Safety and Efficacy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Jewish Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAAVED15A0
Record Dates: First submitted 2016-04-12; First posted 2016-09-29 (Estimated); Results first posted 2022-10-06 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Colistin; Tobramycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard colistin arm (Active Comparator): Subjects initially receive IV colistin 2.5 mg/kg/d divided into three times daily (TID) dosing. Subjects receiving colistin will undergo a 2 day up-titration of dose to an ultimate dose of 4-5 mg/kg/day, for a total treatment of 14 days. The drug is infused over 30 minutes on a TID dosing schedule.
  Interventions: Drug: Colistin
- Modified colistin arm (Active Comparator): Subjects receiving IV colistin undergo a 2 day up-titration to a maximum dose of 5 mg/kg/day, divided into twice daily (BID) dosing, for a total treatment of 14 days. The drug is infused over 30 minutes BID. Steady state plasma concentrations on day 3 of therapy (on 2nd- 3rd dose once at goal dosing) will be measured; specifically, colistin peak (30 minutes after infusion), midpoint (6 hour) and trough (30 minutes prior to next infusion).
  Interventions: Drug: Colistin
- Standard tobramycin arm (Active Comparator): Subjects receive IV tobramycin 8-10 mg/kg/day with once daily dosing for 14 days. Peaks and troughs are drawn with the second dose of tobramycin, and the drug is infused over 30 minutes
  Interventions: Drug: Tobramycin

INTERVENTIONS:
Drug: Colistin
  Arms: Modified colistin arm; Standard colistin arm
Drug: Tobramycin
  Arms: Standard tobramycin arm

SUMMARY:
The purpose of this study is to find the safest and most effective way to administer IV antibiotics to treat acute pulmonary exacerbations (APEs) in patients with cystic fibrosis (CF) that are caused by pathogens, like Pseudomonas aeruginosa. This study will test the safety and effectiveness of two commonly prescribed IV antibiotics: tobramycin and colistin. Though regularly used, not much is known about how these drugs compare with each other in terms of their toxicities, both during short term treatment of an APE and after many treatment courses with these drugs over many years. There are currently no guidelines on the safest and most effective antibiotics to use when treating APEs. We will study kidney function, sputum cultures, and treatment outcomes in patients receiving routine administration of one of these two IV antibiotics. We will also test these outcomes in patients receiving a less frequent dosing schedule for IV colistin. The hope is that this new schedule for IV colistin, which is twice a day and adjusted based on blood and urine tests, will reduce harmful side effects, such as kidney damage, while still being a powerful treatment against CF microbial pathogens.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age at Visit 1.
2. Documentation of CF diagnosis as evidenced by one or more clinical features consistent with the CF phenotype and one or more of the following criteria:

   * Sweat chloride equal or greater than 60 mEq/L by quantitative pilocarpine iontophoresis test.
   * Two well-characterized mutations in the cystic fibrosis transmembrane conductance regulator (CFTR) gene
   * Abnormal nasal potential difference (NPD) as measured by a change in NPD in response to a low chloride solution and isoproterenol of less than -5 mV.
3. Documentation of the presence of an acute pulmonary exacerbation, based on CF Foundation guidelines, as diagnosed by a faculty member of the Denver Adult CF Program.
4. Respiratory culture(s) demonstrating evidence of Pseudomonas aeruginosa or Achromobacter species airway infection.
5. Subject is able to produce sputum, undergo phlebotomy, and provide written consent.
6. The subject's treating physician has determined that they should receive either tobramycin or colistin intravenously as one of the designated agents for their APE treatment. Subjects who are able to receive either tobramycin or colistin as part of their antibiotic regimen will be randomized into one of three arms. If a treating physician deems that a subject cannot receive tobramycin due to vestibular toxicity, ototoxicity or bacterial resistance, the subject will be randomized to either standard or PK-adjusted colistin.

Exclusion Criteria:

1. Concomitant administration of bactrim (due to effects on creatinine).
2. Concomitant administration of inhaled colistin for patients in the colistin PK arm, as this will create inaccuracies in colistin sputum concentration measurements.
3. Patients being treated for B. cepacia, due to colistin resistance by the pathogen.
4. Presence of chronic renal insufficiency, with abnormal baseline creatinine >1.2mg/dL.
5. Presence of a condition or abnormality that in the opinion of the investigator would compromise the safety of the patient or the quality of the data.
6. Inability to perform reproducible spirometry.
7. Inability to expectorate sputum. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-08-26 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2021-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milene Saavedra, MD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Colistin Arm: Subjects initially receive IV colistin 2.5 mg/kg/d divided into three times daily (TID) dosing. Subjects receiving colistin will undergo a 2 day up-titration of dose to an ultimate dose of 4-5 mg/kg/day, for a total treatment of 14 days. The drug is infused over 30 minutes on a TID dosing schedule.
  Colistin
- Modified Colistin Arm: Subjects receiving IV colistin undergo a 2 day up-titration to a maximum dose of 5 mg/kg/day, divided into twice daily (BID) dosing, for a total treatment of 14 days. The drug is infused over 30 minutes BID. Steady state plasma concentrations on day 3 of therapy (on 2nd- 3rd dose once at goal dosing) will be measured; specifically, colistin peak (30 minutes after infusion), midpoint (6 hour) and trough (30 minutes prior to next infusion).
  Colistin
- Standard Tobramycin Arm: Subjects receive IV tobramycin 8-10 mg/kg/day with once daily dosing for 14 days. Peaks and troughs are drawn with the second dose of tobramycin, and the drug is infused over 30 minutes
  Tobramycin
Period: Overall Study
Arm/Group | Standard Colistin Arm | Modified Colistin Arm | Standard Tobramycin Arm
Started | 16 | 10 | 25
Completed | 15 | 10 | 24
Not Completed | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Colistin Arm | Modified Colistin Arm | Standard Tobramycin Arm | Total
Number analyzed (Participants) | 15 | 10 | 24 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 10 | 24 | 49
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (10.6) | 33 (12.3) | 31 (7.2) | 31 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 12 | 31
  Male | 3 | 3 | 12 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 15 | 10 | 24 | 49

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Forced Expiratory Volume at One Second (FEV1) % Predicted Between Study Arms With Acute Pulmonary Exacerbation (APE) Treatment
Description: absolute change in forced expiratory volume at one second (FEV1) % predicted, or percent predicted FEV1, between study arms with acute pulmonary exacerbation (APE) treatment
Time Frame: up to 14 days, from beginning to end of APE treatment
Measure: Mean (Standard Deviation); unit: ppFEV1
Arm/Group | Standard Colistin Arm | Modified Colistin Arm | Standard Tobramycin Arm
Number analyzed (Participants) | 15 | 10 | 24
ppFEV1 | 6.5 (9.5) | 4.4 (3.0) | 4.5 (6.3)

2. Primary Outcome: Rate of Occurrence of the Development of Acute Kidney Injury (AKI) During APE Treatment
Time Frame: up to 14 days, from beginning to end of APE treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Colistin Arm | Modified Colistin Arm | Standard Tobramycin Arm
Number analyzed (Participants) | 15 | 10 | 24
Participants | 1 | 0 | 5

3. Secondary Outcome: Time to Achievement of Steady State With Pharmacokinetic (PK)-Adjusted Colistin Therapy
Time Frame: up to 14 days, from beginning to end of APE treatment
Reporting Status: Not Posted

4. Secondary Outcome: Longitudinal Differences in Exacerbation Rates Between Tobramycin and Colistin Use as Seen in Readmission Rate
Description: time to next admission for exacerbation measured in days when comparing of different antibiotic therapies
Time Frame: from the beginning of APE treatment to 12 months after APE treatment
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Standard Colistin Arm | Modified Colistin Arm | Standard Tobramycin Arm
Number analyzed (Participants) | 15 | 10 | 24
days | 154 (115) | 283 (309) | 241 (184)

5. Secondary Outcome: Differences in Occurrences of Neurotoxicity and Ototoxicity Related Side Effects Between Study Arms as Reported by Treating Physician(s)
Description: absolute occurrences of adverse event rates are being compared between treatment groups using logistic regression, adjusting for age, co-administration of medications such as vancomycin and trimethoprim-sulfamethoxazole, baseline FEV1, admits in the previous year, and diagnosis of CF related diabetes (CFRD) as covariates.
Time Frame: up to 14 days, from beginning to end of APE treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Colistin Arm | Modified Colistin Arm | Standard Tobramycin Arm
Number analyzed (Participants) | 15 | 10 | 24
Participants | 2 | 1 | 1

6. Secondary Outcome: Measurement of Pharmacokinetics of Colistin's Active Metabolites in a Broad CF Population Through Peak, Trough, and Midpoint Blood Draws
Time Frame: up to 14 days, from beginning to end of APE treatment
Reporting Status: Not Posted

7. Secondary Outcome: Comparison of Plasma Pharmacokinetics of Colistin's Active Metabolites With Levels Achieved in the Sputum, in Order to Calculate Epithelial Lining Fluid Concentrations, Through Mass Spectrometry
Time Frame: up to 14 days, from beginning to end of APE treatment
Reporting Status: Not Posted

8. Secondary Outcome: Novel Biomarkers of Nephrotoxic AKI, Prior to Serum Creatinine Increases, Based on Urine Protein:Creatinine Ratios
Time Frame: up to 14 days, from beginning to end of APE treatment
Reporting Status: Not Posted

9. Secondary Outcome: Novel Biomarkers of Nephrotoxic AKI, Prior to Serum Creatinine Increases, Based on the Urine Biomarker Nephrocheck® Point-of-care Assay
Time Frame: up to 14 days, from beginning to end of APE treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 14 days
Description: The total number of participants at risk in each arm of the study represents the number enrolled in each arm of the study, not the total number enrolled. The study arms were not enrolled equally.
Arm/Group | Standard Colistin Arm | Modified Colistin Arm | Standard Tobramycin Arm
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/10 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/10 | 0/24
Other Adverse Events (participants affected / at risk) | 7/15 | 2/10 | 7/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Colistin Arm (N=15) | Modified Colistin Arm (N=10) | Standard Tobramycin Arm (N=24)
Oto- or vestibular toxicity (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Renal toxicity (Renal and urinary disorders) | 1 (1) | 0 (0) | 6 (6)
Oral paresthesias (General disorders) | 4 (4) | 1 (1) | 0 (0)
Headache (General disorders) | 2 (2) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/09/NCT02918409/Prot_SAP_000.pdf
  • Informed Consent Form (2018-12-13): https://cdn.clinicaltrials.gov/large-docs/09/NCT02918409/ICF_001.pdf